CLINICAL TRIAL: NCT00320580
Title: A Randomized, Open-Label, Multicenter Study Comparing the Bleeding Profile of Ortho Evra (Norelgestromin/Ethinyl Estradiol) Continuous Regimen vs. Ortho Evra Cyclic Regimen
Brief Title: An Open-Label Study to Compare the Bleeding Profile of Norelgestromin/Ethinyl Estradiol in an Extended Regimen to Norelgestromin/Ethinyl Estradiol Given in a Traditional Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR008335
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Last update posted 2011-07-01 (Estimated); Status verified 2011-06

CONDITIONS: Metrorrhagia
Keywords: Metrorrhagia; oral contraception; breakthrough bleeding; spotting
MeSH Terms: conditions — Metrorrhagia | interventions — norelgestromin; Ethinyl Estradiol

ARMS (1):
- 001 (Experimental): norelgestromin/ethinyl estradiol
  Interventions: Drug: norelgestromin/ethinyl estradiol

INTERVENTIONS:
Drug: norelgestromin/ethinyl estradiol

SUMMARY:
The purpose of this study is to compare the bleeding profile of norelgestromin/ethinyl estradiol given in an extended continuous regimen to norelgestromin/ethinyl estradiol given in a traditional cyclic regimen

DETAILED DESCRIPTION:
Norelgestromin/ethinyl estradiol is a contraceptive patch shown to be safe and effective for the prevention of pregnancy. The usual treatment regimen is three consecutive seven-day patches followed by one patch-free week. This cyclic method is followed in order to mimic the 28-day menstrual cycle. An extended contraceptive regimen (administration of active hormones for greater than 21 days) of oral contraceptives is a common practice among women wishing to delay or prevent withdrawal bleeding for reasons such as athletic participation or going on vacation. In addition to the convenience of reducing the frequency of withdrawal bleeds, elimination of the hormone-free interval reportedly reduces many menstrually-related symptoms (headaches, pelvic pain, breast tenderness, bloating, swelling) that occur at a greater frequency during the hormone-free interval than during the rest of the cycle. Headache is one of the most common adverse effects associated with hormonal contraceptive use. Studies have demonstrated that headaches were reduced in subjects using extended intervals of active hormone. However, one of the main side effects reported with extended regimens is breakthrough bleeding and/or spotting. Compared to cyclic regimens, extended oral contraceptive use may be associated with an increased incidence of breakthrough bleeding and spotting, especially during the first few months of use. This is a randomized (patients are assigned different treatments based on chance), open-label, multicenter study comparing the bleeding profile of norelgestromin/ethinyl estradiol patch continuous regimen to norelgestromin/ethinyl estradiol patch cyclic regimen. Safety evaluations include adverse event reporting, physical examinations, blood levels, and vital signs. The hypothesis of the study is that norelgestromin/ethinyl estradiol in an extended regimen of 84 days of active hormone would result in fewer days and episodes of bleeding compared to a traditional cyclic regimen of norelgestromin/ethinyl estradiol. Patients receive norelgestromin/ethinyl estradiol patches in a plastic sleeve. In the extended regimen patches will be applied weekly for 12 consecutive weeks followed by one week patch-free and then another three consecutive weeks of weekly patch applications. In the cyclic regimen patches will be applied for four consecutive cycles where each cycle consists of three weekly patch applications followed by one week patch-free. The total duration of treatment period is 112 days for each regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patients in good health as confirmed by medical history
* not pregnant as demonstrated by negative urine pregnancy test
* completed their last term pregnancy at least 42 days prior to Screening and at least one normal menstrual period since last pregnancy
* not lactating
* post-menarcheal and pre-menopausal

Exclusion Criteria:

* History or presence of disorders commonly accepted as contraindications to steroid hormonal therapy including but not limited to the following - active or history of deep vein thrombophlebitis or thromboembolytic disorders or hypercoagulation disorders, cerebral vascular or coronary artery disease, uncontrolled hypertension, or migraines with focal aura, benign or malignant liver tumor which developed during the use of oral contraceptives or estrogen-containing products
* treatment with continuous oral contraception within three months of study
* previous use of contraceptive patch including norelgestromin/ethinyl estradiol
* patients who are amenorrheic (abnormal suppression or absence of menstruation)
* recent history of alcohol or substance abuse
* skin conditions resulting in oily, irritated or damaged skin at potential sites of application

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
The primary efficacy variables are the total number bleeding and/or spotting days during the 84-day reference period and the number of bleeding and/or spotting episodes during the 84-day reference period.

SECONDARY OUTCOMES:
Secondary efficacy variables include the number of breakthrough bleeding and/or spotting days per 28-day interval, the number of breakthrough bleeding days per 28-day interval, time to first bleeding and/or spotting, duration of menses.

CONTACTS AND LOCATIONS:
Overall Officials: McNeil Consumer & Specialty Pharmaceuticals, a Division of Mc Neil-PPC, Inc. Clinical Trial, Study Director — McNeil Consumer & Specialty Pharmaceuticals, a Division of McNeil-PPC, Inc.

REFERENCES:
- [Result] Stewart FH, Kaunitz AM, Laguardia KD, Karvois DL, Fisher AC, Friedman AJ. Extended use of transdermal norelgestromin/ethinyl estradiol: a randomized trial. Obstet Gynecol. 2005 Jun;105(6):1389-96. doi: 10.1097/01.AOG.0000160430.61799.f6. PMID 15932834
- [Result] LaGuardia KD, Fisher AC, Bainbridge JD, LoCoco JM, Friedman AJ. Suppression of estrogen-withdrawal headache with extended transdermal contraception. Fertil Steril. 2005 Jun;83(6):1875-7. doi: 10.1016/j.fertnstert.2004.12.048. PMID 15950671